CLINICAL TRIAL: NCT00940147
Title: Early Indicators for Obstructive Airway Complications After Lung
Brief Title: Early Endoscopic Indicators for OACs After Lung Transplantation: Development of a Novel Mucosal Healing Score
Acronym: OAC
Status: Completed | Type: Observational
Sponsor: Thomas Fuehner (Other)
Responsible Party: Sponsor-Investigator, Thomas Fuehner, Principal Investigator, Hannover Medical School
Organization: Hannover Medical School (Other)
Other Study IDs: 2008_01; OAC_1.0
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Airway Complication Which Require Any Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: patients with OAC, Score finding
- 2: patients without OAC, Score finding

SUMMARY:
Airway complications are a significant cause of morbidity after lung transplantation (LTx). Bronchoscopic evaluation may help to identify risk factors for requiring interventions later.

DETAILED DESCRIPTION:
The investigators evaluated lung transplant recipients prospectively. Adult patients surviving 90 day after LTx will be included. The investigators propose a classification of airway healing based on the endoscopic bronchial appearances at days 7, 14, 21, 90, 180 and 365 after LTx. A score system including mucosal healing, full tissue necrosis (=dehiscence), lose sutures, fibrin plugs, polyps and malacia will be developed (max. score 8 points/date). Endoscopic findings will be correlated with the development of obstructive airway complications (OAC, requiring >1 intervention). Afterwards the new score system will be applied prospectively in the patients.

ELIGIBILITY:
Inclusion Criteria:

* 3 month survivor after LTx
* no OAC

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: LTx 01.2007-05.2009
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoint of this study was any obstructive airway complication (AC) which required desobliterative intervention. | 1 year

SECONDARY OUTCOMES:
secondary endpoint included anastomosis-related death. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- See also: Endoscopic indicators for obstructive airway complications after lung transplantation. — http://www.ncbi.nlm.nih.gov/pubmed/20885336